CLINICAL TRIAL: NCT03062020
Title: New Tool to Predict Risk of Spontaneous Preterm Birth in Asymptomatic High-risk Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Montse Palacio, Medical Doctor. Physician Doctor. Senior consultant, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HCB/2016/0552
Record Dates: First submitted 2016-11-29; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: PreTerm Birth
Keywords: Preterm Birth; Asymptomatic high-risk women; QUIPP; Quantitative fetal fibronectin; Cervical length
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: QUIPP tool arm (Experimental): In this group, QUIPP tool will be used to select and manage patients attending our PBPC: high-risk patients will be followed-up in our PBPC and low-risk patients will be discharged from PBPC and managed in a low-risk unit.
  Interventions: Device: QUIPP
- Control group: no QUIPP tool arm (No Intervention): Women will be managed according to current clinical practice.

INTERVENTIONS:
Device: QUIPP — Information required by QUIPP tool will be introduced ( obstetrical history, cervical length and quantitative fetal fibronectin value) and a percentage of risk of preterm birth will be given. Women with a high-risk value will be managed in Preterm Birth Prevention Clinic and women with low-risk value will be followed-up in a low-risk unit.
  Arms: Intervention group: QUIPP tool arm

SUMMARY:
The QUIPP tool integrates information of obstetrical history, quantitative fetal fibronectin (qfFN) and cervical length to predict the risk of sPTB in asymptomatic high-risk women.

The aim of this study is to evaluate the QUIPP tool in our setting in order to optimize the management of women at high risk for sPTB and to validate in a randomized clinical trial, whether the use of QUIPP improves efficiently the management of our asymptomatic high-risk women when it is compared with the current clinical management.

Design: Randomized controlled trial. Inclusion criteria: Asymptomatic singleton pregnancies 18,0-22,6 weeks at high-risk for sPTB. Sample size: According to a non-inferiority analysis, 129 pregnant women will be needed for each arm.

Methodology: Patient selection and who consent to participate in the study will be randomized into two arms: a) Intervention group: QUIPP tool will be used to select and manage patients attending our PBPC: high-risk patients will be followed-up in our PBPC and low-risk patients will be discharged from PBPC and managed in a low-risk unit. b) Control group: Women will be managed according to current clinical practice.

Main Outcome: sPTB <34,0 and <37,0 weeks of gestation. Secondary Outcomes: Pregnancy outcomes and a neonatal composite morbidity. Expected Results: Perinatal outcomes are similar in the intervention and control group although the intervention group using the QUIPP tool required less medical resources.

DETAILED DESCRIPTION:
Preterm birth (PTB) is a leading cause of perinatal morbidity and mortality. Women at high-risk of preterm birth are those with a previous spontaneous preterm birth (sPTB) or preterm premature rupture of membranes before 35 weeks of gestation, uterine malformation, surgery on uterine cervix or a short cervical length; these women have a global risk of PTB about 30% but still 75%-85% of these women will deliver at term without any intervention.

The availability of a specialized Preterm Birth Prevention Clinic (PBPC) is relevant for the management of these high-risk pregnant women and it results in a reduction in the risk of recurrent sPTB, pregnancy prolongation and a reduction in the rate of major neonatal morbidity. However, it implies higher outpatient care costs as well as trained personnel and intensive follow-up management even for those women not destined to deliver preterm QUIPP is a free smartphone application that integrates the obstetrical history of high-risk women, the cervical length and the value of quantitative fetal fibronectin to predict the risk of preterm birth. QUIPP will determinate the risk of preterm birth in these high-risk women.

Patients will be randomized in two groups: Intervention group (QUIPP tool arm): QUIPP tool is applied and patients with a high-risk result will be follow-up in a high-risk unit (PBPC) and patients with a low-risk value will be managed in a low-risk unit. Control group (no QUIPP tool arm): current management in a PBPC will be applied.

The use of QUIPP will allow determining which asymptomatic pregnancies with risk factors for sPTB will deliver preterm. Furthermore, we expect to provide the non-specialized clinician with an objective, useful, accurate and efficient tool to manage these women with same pregnancy and neonatal outcomes and using less resource.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Asymptomatic singleton pregnancies, with at least one of the following: Previous spontaneous preterm delivery or a preterm premature rupture of membranes ≤ 346 weeks of gestation, Previous spontaneous second trimester miscarriage, Previous surgery on uterine cervix, Incidental finding of cervical length less than 25mm, Uterine malformations.
* Able to sign informed consent form.

Exclusion Criteria:

* Multiple pregnancies.
* Congenital, chromosomal abnormalities or stillbirth in current pregnancy.
* No patient consent to participate in the study
* Women with an obstetrical history of iatrogenic preterm birth indicated for maternal or fetal conditions.
* Symptomatic high-risk women or preterm prelabor rupture of membranes in current pregnancy.
* Pregnant women with an indication of prophylactic cervical cerclage due to her own obstetrical history.
* Pregnant women with a short cervix detected by ultrasound and with an indication to perform a cervical cerclage, prior to study inclusion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2016-11-16 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Spontaneous preterm birth before 34.0 and 37.0 weeks of gestation | 3.5 years
  Delivery < 34.0 and <37.0 weeks of gestation ( Yes/No )

SECONDARY OUTCOMES:
Gestational age at delivery | 3,5 years
  Weeks and days at the moment of delivery
Hospital admission due to sPTB or PPROM | 3.5 years
  Number of hospital admission due to a spontaneous preterm labor or a preterm premature rupture of membranes
Emergency department visits due to uterine contractions | 3.5 years
  Number of emergency department visits
Clinical chorioamnionitis | 3.5 years
  Fever ( >37.8 ºC) and maternal tachycardia ( >100 beats per minute) and /or fetal tachycardia ( >160 beats per minute) and/or maternal leukocytosis ( >15000 leukocites/mm3) and/or uterine contractions and/or malodorous leukorrhea
Maternal mortality | 3.5 years
  Maternal death (Yes/No)
5 min APGAR score <7 | 3.5 years
  APGAR test less than 7 at the 5 minuts after birth
umbilical artery pH at delivery <7.1 | 3.5 years
  pH artery value less than 7.1
NCIU admission | 3.5 years
  Admission in a neonatal intensive care unit ( Yes/No)
Need for respiratory support | 3.5 years
  Administration of respiratory support during the NCIU stay.
Respiratory distress syndrome | 3.5 years
  Breathing disorder ( Yes /No)
Intraventricular haemorrhage | 3.5 years
  Severe intraventricular haemorrhage grade III/IV
Necrotizing enterocolitis | 3.5 years
  Intestinal necrosis in the newborn ( Yes/No)
Neonatal sepsis | 3.5 years
  Blood infection of the newborn (Yes/No)
Neonatal mortality | 3.5 years
  neonatal death

CONTACTS AND LOCATIONS:
Overall Officials: Núria Lorente, M.D, Principal Investigator — BCNatal | Barcelona Center for Maternal Fetal and Neonatal Medicine | Hospital Clínic - Hospital Sant Joan de Déu
Locations (2):
- Spain (2):
  - Hospital Clínic Barcelona ( Maternitat), Barcelona, Barcelona
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtzman J, Chandiramani M, Briley A, Poston L, Das A, Shennan A. Quantitative fetal fibronectin screening in asymptomatic high-risk patients and the spectrum of risk for recurrent preterm delivery. Am J Obstet Gynecol. 2009 Mar;200(3):263.e1-6. doi: 10.1016/j.ajog.2009.01.018. PMID 19254585
- [Background] Abbott DS, Hezelgrave NL, Seed PT, Norman JE, David AL, Bennett PR, Girling JC, Chandirimani M, Stock SJ, Carter J, Cate R, Kurtzman J, Tribe RM, Shennan AH. Quantitative fetal fibronectin to predict preterm birth in asymptomatic women at high risk. Obstet Gynecol. 2015 May;125(5):1168-1176. doi: 10.1097/AOG.0000000000000754. PMID 25932845
- [Background] Kuhrt K, Smout E, Hezelgrave N, Seed PT, Carter J, Shennan AH. Development and validation of a tool incorporating cervical length and quantitative fetal fibronectin to predict spontaneous preterm birth in asymptomatic high-risk women. Ultrasound Obstet Gynecol. 2016 Jan;47(1):104-9. doi: 10.1002/uog.14865. PMID 25846437